CLINICAL TRIAL: NCT05270031
Title: A Phase 3 Randomized Controlled Clinical Trial: Balloon Dilation Treatment of the Eustachian Tube Using an Endovascular Balloon
Brief Title: Balloon Dilation of the Eustachian Tube
Acronym: BDET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3156
Record Dates: First submitted 2021-09-21; First posted 2022-03-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Intervention Model Description: Cross Over after 3 months possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eustachian tube dilation (Experimental): Surgical Eustachian tube dilation in general anaesthesia
  Interventions: Device: Balloon dilation of the eustachian tube
- Control Group (No Intervention): nasal saline spray

INTERVENTIONS:
Device: Balloon dilation of the eustachian tube — Balloon dilation of the eustachian tube
  Arms: Eustachian tube dilation

SUMMARY:
In this study, patients with dysfunction of the eustachian tube will be included. They will be randomized to one of two treatment groups.

1. balloon dilation of the eustachian tube or
2. nasal saline Patients will undergo follow-up for one year and will be able to crossover to the treatment arm after three months

DETAILED DESCRIPTION:
Patients will eustachian tube dysfunction will be asked to participate in the study.

They will be randomized to one of two groups

group 1 - surgical dilation of the eustachian tube in general anaesthesia

group 2 - daily nasal saline spray, twice a day

Regular Follow up with Tympanogram and Questionnaire

After three months patient in the control group (nasal saline) can switch in the intervention group.

Eustachian tube dilation will be carried out with a Health Canada and FDA approved device, usually used for endovascular balloon dilation. It has the same size and pressure properties as the eustachian tube dilation device and has shown a good safety profile in a previous preclinical and clinical pilot study.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old (of both sexes)
* Diagnosed with persistent obstructive eustachian tube dysfunction (OETD) for at least 3 months prior to enrolment uni- and/or bilateral

Diagnosis (both required):

i. Persistent OETD symptoms assessed by Eustachian Tube Dysfunction Questionnaire (ETDQ-7) with overall score of ≥3 (moderate to severe symptoms) for 3 months or more prior to enrollment.

ii. Refractory to medical therapy (minimum of 4 weeks of daily intranasal steroid spray or one completed course of an oral steroid within 3 months before study enrollment).

Exclusion Criteria:

* Patulous eustachian tube
* Prior eustachian tube intervention
* Presence of myringotomy ventilation tube or a tympanic membrane perforation
* Active chronic or acute otitis media
* Chronic otitis media with cholesteatoma
* Fluctuating sensorineural hearing loss or Meniere's disease
* Chronic rhinosinusitis, allergies, or reflux disease not controlled with medication
* History of head or neck surgery within 3 months
* Prior radiation to the head and neck
* Active temporomandibular joint disorders
* Cleft palate or Craniofacial syndrome
* Cystic fibrosis or Ciliary dysmotility syndrome or Systemic immunodeficiencies
* Active acute upper respiratory infection
* Nasal endoscopy with evidence of anatomic conditions that would prevent transnasal access to the Eustachian tube
* CT temporal bone scan with evidence of carotid artery dehiscence, superior semicircular canal dehiscence, or extrinsic eustachian tube compression
* Patient unable to follow protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Otoscopy, Normal, Retracted or Middle ear effusion | 6 weeks
  Microscopic evaluation of tympanic membrane
Otoscopy, Normal, Retracted or Middle ear effusion | 3 motnths
  Microscopic evaluation of tympanic membrane
Otoscopy, Normal, Retracted or Middle ear effusion | 6 months
  Microscopic evaluation of tympanic membrane
Otoscopy, Normal, Retracted or Middle ear effusion | 12 months
  Microscopic evaluation of tympanic membrane

SECONDARY OUTCOMES:
Valsalva maneuver -positive or negative | 6 weeks
  Subjective effectiveness of Valsalva maneuver
Valsalva maneuver -positive or negative | 3 months
  Subjective effectiveness of Valsalva maneuver
Valsalva maneuver -positive or negative | 6 months
  Subjective effectiveness of Valsalva maneuver
Valsalva maneuver -positive or negative | 12 months
  Subjective effectiveness of Valsalva maneuver
Tympanogram | 3 months
  Measurement with tympanometer
Tympanogram | 6 months
  Measurement with tympanometer
Tympanogram | 12 months
  Measurement with tympanometer
ETDQ-7 (eustachian tube dilation questionnaire - seven) | 6 weeks
  Questionnaire
ETDQ-7 (eustachian tube dilation questionnaire - seven) | 3 months
  Questionnaire
ETDQ-7 (eustachian tube dilation questionnaire - seven) | 6 months
  Questionnaire
ETDQ-7 (eustachian tube dilation questionnaire - seven) | 12 months
  Questionnaire
HUI (Health utility index) | 6 weeks
  Questionnaire
HUI (Health utility index) | 3 months
  Questionnaire
HUI (Health utility index) | 6 months
  Questionnaire
HUI (Health utility index) | 12 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Trung N Le, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607